CLINICAL TRIAL: NCT06380803
Title: Surgical Skill Labs for Robotic Mastectomy Using Cadaver And Porcine Models and Educational Program Using a Surgical Guide by Artificial Intelligence
Brief Title: Surgical Skill Labs for Robotic Mastectomy and Educational Program Using a Surgical Guide by Artificial Intelligence
Acronym: ROMCAPO+AI
Status: Recruiting | Type: Observational
Sponsor: Severance Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Hyung Seok Park, MD, PhD, Professor, Department of Surgery, Principal Investigator, Severance Hospital
Other Study IDs: 4-2020-1385
Record Dates: First submitted 2024-02-28; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Breast Neoplasms; Surgery; Educational Problems; Surgical Procedure, Unspecified
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: A educational program — A educational program using cadaver or porcine models for robotic brest surgery

SUMMARY:
The goal of this prospective study is to investigate the satisfaction, NASA-Task Load Index (TLX), and surgical proficiency of a robotic breast surgery education program using cadaver or porcine models, as well as to develop an AI-based surgical guide for utilization within the educational program in trainees for robotic breast surgery.

The main question[s]it aims to evaluate :

* Satisfaction questionnaire of a educational program
* NASA-TLX of a educational program
* global evaluative assessment of robotic skills (GEARS) of a robotic breast surgery for surgical proficiency

Participants will participate the educational program and fill out a satisfaction questionnaire and NASA-TLX.

The tutor evaluates GEARS for 15 minutes at the beginning and end of training.

After the development of the surgical guide based on AI, researchers will compare a training group with or without surgical guide to see the effect of the surgical guide.

DETAILED DESCRIPTION:
The goal of this prospective study is to investigate the satisfaction, NASA-Task Load Index (TLX), and surgical proficiency of a robotic breast surgery education program using cadaver or porcine models, as well as to develop an AI-based surgical guide for utilization within the educational program in trainees for robotic breast surgery.

The main aims to evaluate the satisfaction questionnaire, NASA-TLX of a educational program, and global evaluative assessment of robotic skills (GEARS) of a robotic breast surgery for surgical proficiency.

Participants will participate the educational program and fill out a satisfaction questionnaire and NASA-TLX. The tutor evaluates GEARS for 15 minutes at the beginning and end of training. After the development of the surgical guide based on AI, researchers will compare a training group with or without surgical guide to see the effect of the surgical guide.

The inclusion criteria is as below; a breast surgeon who completed the basic dry lab for surgical robot platform before the educational program and a trainee who signed a informed consent.

The exclusion criteria is as below; a trainee who did not sign a informed consent and a trainees judged by the researcher to be inappropriate for participation in this study.

The estimated participants is at least 64.

This study will present the descriptive statistics on the collected data of the satisfaction questionnaire, NASA-TLX, and GEARS results. Categorial variables will be examined by the chi-square test or Fisher's exact test. Continuous variables will be examined by t-test or M-W test if needed. Additionally, binary regression test will be tested for multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* A breast surgeon who completed the basic dry lab for surgical robot platform before the educational program
* A trainee who signed a informed consent

Exclusion Criteria:

* A trainee who did not sign a informed consent
* A trainees judged by the researcher to be inappropriate for participation in this study

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: any breast surgeon who participate a educational program using cadavers or porcine models for robotic breast surgery
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2025-01-26 (Estimated); Study Completion 2025-01-26 (Estimated)

PRIMARY OUTCOMES:
Satisfaction questionnaire of a educational program | 1 day
  (grading scale: 1-insufficient/inadequate; 2-reasonable/adequate; 3-sufficient; 4-good; 5-very good.)
  Participants' perceived goals for attending the course:
  1. Met expectations in knowledge (theory),
  2. met expectations in skill practice,
  3. met knowledge requirements in theory,
  4. met the essentials in skills development,
  5. developed participants at skills performance.
     Teaching/learning environment:
  6. ambience of the laboratory,
  7. structure of the session,
  8. pace of the session,
  9. mix explanation/opportunity to practise,
  10. environment & content valuable for understanding,
  11. participants' involvement,
  12. development of participants' interest in the skills,
  13. training adequacy.
      Teaching staff performance:
  14. Relationship with participants,
  15. enthusiasm for teaching,
  16. encouragement of participants' participation,
  17. clear explanations,
  18. clear demonstration of each component of the skill,
  19. 'feedback'
NASA-Task Load index of a educational program | 1 day
  Hart and Staveland's NASA Task Load Index method assesses work load on five 7-point scales. Increments of high, medium and low estimates for each point result in 21 gradations on the scales. (grading scale: 1- very low; 21-very high.)
  1. Mental Demand: How mentally demanding was the task?
  2. Physical Demand: How physically demanding was the task?
  3. Temporal Demand: How hurried or rushed was the pace of the task?
  4. Performance: How successful were participants in accomplishing what participants were asked to do?
  5. Effort: How hard did participants have to work to accomplish participants' level of performance?
  6. Frustration: How insecure, discouraged, irritated, stressed, and annoyed were participants?
Global Evaluative Assessment of Robotic Skills of a robotic breast surgery for surgical proficiency | 1 day
  The Global Evaluative Assessment of Robotic Skills assessment involves conducting an initial evaluation for 15 minutes at the beginning of the education session and a second evaluation for 15 minutes before the end of the session, evaluating the improvement in skill level based on the difference between the two evaluation scores.
  (grading scale: 1- very poor; 2 - poor; 3 - average; 4 - good; 5 - excellent.)
  1. Depth perception :
  2. bimanual dexterity:
  3. efficiency:
  4. force sensitivity:
  5. autonomy:
  6. robotic control:

SECONDARY OUTCOMES:
The comparison of satisfaction questionnaire of a educational program between the group with the surgical guide and without the surgical guide | through study completion, an average of 4 year
  The investigators will conduct descriptive statistical analysis of satisfaction questionnaire of a educational program. When conducting subgroup analysis within all subjects between the group with the surgical guide group and the group without the surgical guide, univariate and multivariate analysis will be performed, and the analysis will be conducted in accordance with general statistical processing.
  The detailed scale of the satisfaction questionnaire of a educational program is the same as the primary outcome measures.
The comparison of NASA-Task Load index of a educational program between the group with the surgical guide and without the surgical guide | through study completion, an average of 4 year
  The investigators will conduct descriptive statistical analysis of NASA-Task Load index of a educational program. When conducting subgroup analysis within all subjects between the group with the surgical guide group and the group without the surgical guide, univariate and multivariate analysis will be performed, and the analysis will be conducted in accordance with general statistical processing.
  The detailed scale of NASA-Task Load index of a educational program is the same as the primary outcome measures.
The comparison of Global Evaluative Assessment of Robotic Skills of a robotic breast surgery for surgical proficiency between the group with the surgical guide and without the surgical guide | through study completion, an average of 4 year
  The investigators will conduct descriptive statistical analysis of Global Evaluative Assessment of Robotic Skills of a robotic breast surgery for surgical proficiency. When conducting subgroup analysis within all subjects between the group with the surgical guide group and the group without the surgical guide, univariate and multivariate analysis will be performed, and the analysis will be conducted in accordance with general statistical processing.
  The detailed scale of Global Evaluative Assessment of Robotic Skills of a robotic breast surgery for surgical proficiency is the same as the primary outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Hyung Seok Park, MD, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] da Costa PM, Santos J, Maio R, Santos A, Paredes F. The role of a basic surgical skills laboratory as viewed by medical students (6th year). Med Teach. 2001 Mar;23(2):176-180. doi: 10.1080/01421590120036565. PMID 11371295
- [Background] Goh AC, Goldfarb DW, Sander JC, Miles BJ, Dunkin BJ. Global evaluative assessment of robotic skills: validation of a clinical assessment tool to measure robotic surgical skills. J Urol. 2012 Jan;187(1):247-52. doi: 10.1016/j.juro.2011.09.032. Epub 2011 Nov 17. PMID 22099993
- [Background] Wilson MR, Poolton JM, Malhotra N, Ngo K, Bright E, Masters RS. Development and validation of a surgical workload measure: the surgery task load index (SURG-TLX). World J Surg. 2011 Sep;35(9):1961-9. doi: 10.1007/s00268-011-1141-4. PMID 21597890